CLINICAL TRIAL: NCT06047158
Title: Effects of Omega-3 Fish Oil Fat Emulsion on Rehabilitation and Immune Function After Radical Surgery Combined With Intraperitoneal Hyperthermic Infusion Chemotherapy in Patients With Locally Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: RCEOFOITP
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Fish Oils; Perfusion; Complications; Stomach Neoplasms; Nutrition Aspect of Cancer; Chemotherapy Effect; Immunisation Reaction
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fish oil group: The patients in this group were treated with omega-3 fish oil fat emulsion at a dose of 100ml/ per person per day for 5 days and added to a three-liter bag (containing water, glucose, amino acids, sodium chloride, vitamins, etc.) except fish oil.
  Drug introduction:
  Full name: omega-3 fish oil fat emulsion. Common name: Juventus. Specification: 100ml / 10g
  Interventions: Drug: Omega-3 fish oil fat emulsion
- Non-fish oil group: Do not use omega-3 fish oil fat emulsion (no omega-3 fish oil fat emulsion is added to the three-liter bag, other substances are the same)

INTERVENTIONS:
Drug: Omega-3 fish oil fat emulsion — Use omega-3 fish oil fat emulsion
  Groups: Fish oil group

SUMMARY:
The purpose of this study was to investigate the effects of omega-3 fish oil fat emulsion on peripheral blood C-reactive protein, total lymphocyte count, plasma albumin and immune function after radical surgery combined with intraperitoneal hyperthermic perfusion chemotherapy in patients with locally advanced gastric cancer. at the same time, to explore the effects of omega-3 fish oil fat emulsion on complications, length of stay and total cost of hospitalization.

The main question it aims to answer is whether the use of omega-3 fish oil fat emulsion can improve patients' immunity, speed up recovery and reduce costs.

Participants will comprehensively collect patient-related baseline data, including sex, age, BMI, ASA grade, tumor location, histological grade, pathological tumor type, pTNM stage (AJCC cancer stage 8), and perilymphatic vascular / nerve infiltration.

Immune function evaluation related index: peripheral blood lymphocyte count. Plasma albumin concentration, C-reactive protein, postoperative infectious complications, length of stay and cost of hospitalization.

Finally, statistical analysis software was used to analyze the differences between the two groups, evaluate the above indicators and draw mutual conclusions.

DETAILED DESCRIPTION:
The research process is as follows:

1. Select patients in the group according to the inclusion and exclusion criteria.
2. The patient signed the informed consent form
3. His system was used to collect patient data, including human-related baseline data, including sex, age, BMI, ASA grade, tumor location, histological grade, pathological tumor type, pTNM stage (AJCC cancer stage 8th edition), lymphatic vascular / nerve infiltration. Immune function evaluation related index: peripheral blood lymphocyte count. Plasma albumin concentration, C-reactive protein, postoperative infectious complications, length of stay and cost of hospitalization.
4. Using statistical software (SPSS) to judge the statistical difference.
5. It is concluded that the use value of omega-3 fish oil fat emulsion (Ewing) is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The age is 18 to 75 years old.
* For advanced gastric cancer, according to the TNM staging specified by the 8th edition AJCC, the clinical staging or EUS staging is above T2. There is no distant metastasis before operation, and the tumor does not directly invade the surrounding organs (liver, pancreas, spleen and transverse mesocolon, etc.).
* There is no obvious contraindication to surgery.
* The preoperative physical status score of Eastern American Cancer Cooperation (ECOG) was 0 or 1.
* The preoperative ASA grade was grade Ⅰ-Ⅲ.
* No previous history of gastric surgery, no history of other malignant tumors.
* After explaining the nature and purpose of the study, agree to sign an informed consent form, give voluntary consent to participate in the study, and comply with the requirements of the study.

Exclusion Criteria:

* Radiotherapy or chemotherapy before operation.
* Use of immunosuppressants such as hormones within 3 months before treatment.
* Preoperative anemia (hemoglobin < 90g/L) and severe hypoalbuminemia (albumin < 30g/L).
* With severe heart and lung and other important organ dysfunction.
* More serious metabolic and immune diseases, such as hyperthyroidism, poor blood glucose control in diabetes, obesity, hyperlipidemia (triglyceride > 3mmol/L, total bile solid > 6.2mmol/L).
* Severe infection before operation.
* With complete intestinal obstruction, intestinal perforation and intestinal necrosis.
* During the operation, it was found that radical operation could not be performed or combined organ resection was needed.
* Operation time > 6 hours, intraoperative bleeding > 400ml

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population were patients with advanced gastric cancer who had received surgical treatment. According to the wishes of the patients, they chose whether to use omega-3 fish oil fat emulsion and were assigned to different groups to observe the effect.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Immune related index | one week
  Peripheral blood lymphocyte count
Immune related index | one week
  Plasma albumin concentration
Immune related index | one week
  C-reactive protein concentration
Immune related index | one week
  Postoperative infectious complications

SECONDARY OUTCOMES:
Hospitalization related | From the first day after operation to discharge, up to 30 days.
  Hospitalization time
Hospitalization related | From the first day after operation to discharge, up to 30 days.
  Hospitalization expenses

CONTACTS AND LOCATIONS:
Locations (1):
- Ruiqing Liu, Qingdao, Shandong, China